CLINICAL TRIAL: NCT06817187
Title: A Single Center, Randomized, Open Label, Controlled Clinical Study to Evaluate the Mutual Influence of Combined Administration of 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular Pertussis (Component) Combined Vaccine (Adsorbed)
Brief Title: Clinical Study on the Combined Administration of 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus, Pertussis Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 201904003
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Streptococcus Pneumoniae Infections
Keywords: 15-valent pneumococcal conjugate vaccine; Diphtheria, Tetanus, Pertussis Vaccine
MeSH Terms: conditions — Pneumococcal Infections; Diphtheria; Tetanus | interventions — Tetanus Toxoid; Elements; Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- P+DTP group (Experimental): 370 infants aged 3 months were enrolled in this group.
  Interventions: Biological: 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed)
- P-DTP group (Experimental): 370 infants aged 3 months were enrolled in this group.
  Interventions: Biological: Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed)
- DTP group (Active Comparator): 370 infants aged 3 months were enrolled in this group.
  Interventions: Biological: 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed)

INTERVENTIONS:
Biological: 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed) — Administer 0.5ml of 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed) separately at different locations upon enrollment. Both vaccine were immunized according to the 0, 1, and 2 month procedures (calculated as 30 days per month).
  Arms: DTP group
Biological: 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed) — Vaccination with 15-Valent Pneumococcal Conjugate Vaccine with a 7-day interval (+15 day window period) followed by vaccination with Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed). Both vaccine were immunized according to the 0, 1, and 2 month procedures (calculated as 30 days per month).
  Arms: P+DTP group
Biological: Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed) — Only administer the Diphtheria, Tetanus and Acellular pertussis (Component) Combined Vaccine (Adsorbed) and according to the 0, 1, and 2 month procedures (calculated as 30 days per month).
  Arms: P-DTP group

SUMMARY:
This clinical study aims to evaluate the mutual influence of combined administration of 15-Valent Pneumococcal Conjugate Vaccine and Diphtheria, Tetanus, Pertussis Vaccine in the target population

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 3 months (90-119 days old), full-term (37-42 weeks pregnant), with a birth weight of ≥ 2.5kg;
* The legal guardian provides informed consent and signs the informed consent form;
* The legal guardian agrees to comply with the requirements of the clinical research protocol, is willing to accept a follow-up of 10 months, and has the ability to use thermometers, scales, and fill out diary cards; 4) Have not received pneumococcal vaccine or pertussis vaccine, and have no history of receiving other live vaccines in the past 14 days or non live vaccines in the past 7 days; 5) Underarm temperature ≤ 37.0 ℃.

Exclusion Criteria:

* A history of invasive diseases caused by Streptococcus pneumoniae that has been confirmed through cultivation;
* Known to be allergic to any component of the experimental vaccine, especially those allergic to diphtheria toxoid, or those who previously have a fever of 39.5 ℃ or above after receiving vaccine;
* History or family history of seizures, epilepsy, encephalopathy, and mental illness;
* Infants born with abnormal labor processes (difficult labor, instrumental delivery) or with a history of asphyxia or neurological organ damage;
* A history of confirmed thrombocytopenia or other coagulation disorders may result in contraindications for subcutaneous injection;
* Injecting human normal immunoglobulin after birth;
* Known or suspected immunological dysfunction, receiving immunosuppressive therapy (radiation therapy, chemotherapy, corticosteroids, antimetabolites, cytotoxic drugs), such as continuous treatment with systemic corticosteroids (prednisone or similar drugs) for ≥ 14 days, human immunodeficiency virus (HIV) infection, etc;
* Having congenital malformations, severe malnutrition, developmental disorders, and genetic defects (such as favism);
* Currently suffering from serious chronic diseases, infectious diseases, active infections, liver diseases, kidney diseases, cardiovascular diseases, and malignant tumors;
* Severe asthma;
* Systemic rash, skin ringworm, skin suppuration or blisters;
* Currently or planning to participate in clinical trials of other drugs in the near future; Researchers believe that any situation that may affect the evaluation of the study.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1110 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Antibody positive conversion rate | 30 days after full vaccination
  The positive conversion rates of diphtheria antibody (anti-D), tetanus antibody (anti-T), pertussis toxin antibody (anti-PT), and pertussis filamentous hemagglutinin antibody (anti-FHA) in P+DTP, P-DTP, and DTP groups，respectively.

SECONDARY OUTCOMES:
AEs within 0-30 minutes after vaccination | 0-30 minutes after vaccination
  The occurrence of all adverse events within 0-30 minutes after each dose of vaccination
Solicited AEs within 0-7 days after vaccination | 0-7 days after vaccination
  The occurrence of all solicited adverse events within 0-7 days after each dose of vaccination
Unsolicited AEs within 0-30 days after vaccination | 0-30 days after vaccination
  The occurrence of all unsolicited adverse events within 0-30 days after each dose of vaccination.
SAE within 0-6 months after primary immunization | 0-6 months after primary immunization
  The occurrence of all serious adverse events within 0-6 months after primary immunization.
Positive rate of IgG antibodies | 30 days after full vaccination
  Positive rate of susceptible individuals with 15 serotype specific pneumococcal IgG antibodies (percentage of subjects with antibody concentration ≥ 0.35 μ g/ml)
GMC of IgG antibody | 30 days after full vaccination
  GMC of IgG antibody against 15 serotype specific pneumococcal.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Doctor, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei, China